CLINICAL TRIAL: NCT06083077
Title: Effect of Chest and Abdominal Wall Strapping on Ventilation and Work of Breathing in Infants With Severe Bronchiolitis: a Physiological Study
Brief Title: Chest and Abdominal Wall Strapping in Infant With Bronchiolitis
Acronym: WRAPITIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: As the epidemiology of bronchioles has changed over the last two winters with the introduction of beyfortus, we have few eligible patients.
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL23_0821
Record Dates: First submitted 2023-09-25; First posted 2023-10-13 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Bronchiolitis
Keywords: Bronchiolitis; Work of breathing; Non-invasive ventilation; Infant
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: Infant will be recorded successively in 6 conditions (10 min each) :
  * Without chest wall strapping at PEEP (Positive End Expiratory Pressure) 0 and PEEP 7
  * With chest wall strapping at PEEP 0 and PEEP 7
  * again without chest wall strapping at PEEP 0 and PEEP 7.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Infant < 6 months with severe bronchiolitis (Experimental): Infant will be recorded successively in 6 conditions (10 min each) :
  * Without chest wall strapping at PEEP 0 and PEEP 7
  * With chest wall strapping at PEEP 0 and PEEP 7
  * again without chest wall strapping at PEEP 0 and PEEP 7.
  Interventions: Other: Chest wall strapping

INTERVENTIONS:
Other: Chest wall strapping — An elastic band (6 cm wide) is placed around the lower part of the chest wall (at the junction of the chest and abdomen) to tighten the chest wall for 10 min at PEEP 7 cmH2O and 10 min without PEEP

SUMMARY:
Bronchiolitis is the most common cause of admission to the Paediatric Intensive Care Unit (PICU) for respiratory distress.

The care of an infant with severe bronchiolitis is mainly based on symptomatic treatment (nutritional and respiratory support). The lower part of an infant's chest is larger than that of an older child, which can flatten the diaphragm, especially in obstructive disease with air trapping. Strapping the lower part (at the junction of the chest and abdomen) may provide a better condition for diaphragmatic contraction. Based on respiratory mechanics in infants and physiological studies in adults, investigators hypothesise that chest wall strapping may improve the ventilation and the diaphragmatic contraction.

Infant < 6 month with severe bronchiolitis admitted to the PICU will be recorded in 4 conditions with or without chest wall strapping and with a Continuous Positive Airway Pressure (CPAP) at 7 cmH2O or without CPAP. Physiological parameters (including work of breathing, respiratory parameters, distribution of ventilation) will be recorded and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Infant < 6 months
* Admitted to the PICU for less than 48 hours
* With a diagnosis of bronchiolitis
* With a respiratory distress sign (mWCAS ≥ 3) and non-invasive ventilatory support
* With a naso or oro gastric tube for feeding
* With written informed consent from parents or legal guardians

Exclusion Criteria:

* Infants with severe bronchopulmonary disease, severe laryngomalacia, neuromuscular disease, bone disease, cyanotic heart disease
* Contraindication to the use of a gastric tube
* recent abdominal or thoracic surgery
* investigator able to perform physiological recording not available
* Patient who is not affiliated (or does not benefit from) to a national social security system

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Esophagal product time pressure | 1 hour
  Average over 100 consecutive cycles of esophageal product time pressure value

SECONDARY OUTCOMES:
Diaphragmatic product time pressure | 1 hour
  Average over 100 consecutive cycles of diaphragmatic product time pressure value
Esophagal and diaphragmatic swing | 1 hour
  Mean on 100 breaths of the amplitude (maximum value -minimum value) of the esophageal pressure (cmH2O) and gastric pressure (cmH2O)
Distribution of ventilation : center of ventilation | 1 hour
  Mean over 1 minute of the center of the ventilation (%). Center of ventilation represents the average of the dorsal-ventral distribution of tidal variation using Electrical Impedance Tomography (values >50% indicating that the center of ventilation is located in the ventral part of the chest)
End expiratory lung volume | 1 hour
  Average over 1 minute of the end expiratory lung impedance
Time ratio | 1 hour
  average over 100 consecutive cycles of inspiratory to aspiratory time ratio
modified wood asthma score (mWCAS) | 1 hour
  Value of the modified wood asthma score at the end of the recording period in each condition.
  Minimal value 0 and maximal value 10. A score ≥ 3 mean a moderate-to-severe respiratory distress.
TcPCO2 | 1 hour
  Average of the transcutaneous CO2 (carbon dioxide) partial over 1 minute
EDIN scale (Newborn Pain and Discomfort Scale) | 1 hour
  Value of the EDIN score at the end of the recording period in each condition. Minimal value 0 and maximal value 15. EDIN scores > 6 are considered expression of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Réanimation pédiatrique, Bron, France

IPD SHARING:
Plan to Share IPD: No